CLINICAL TRIAL: NCT00868517
Title: The Effect of Acupuncture on PTSD-Related Insomnia
Brief Title: Examining the Effect of Acupuncture on Sleep Difficulties Related to Post Traumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NRI 08-121
Record Dates: First submitted 2009-03-23; First posted 2009-03-25 (Estimated); Results first posted 2014-11-17 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2014-09

CONDITIONS: Stress Disorders, Post-Traumatic; Sleep Initiation and Maintenance Disorders
Keywords: Veterans; Operation Iraqi Freedom; Operation Enduring Freedom; Combat Disorders; Acupuncture; Complementary Therapies
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sleep Initiation and Maintenance Disorders; Combat Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- True Group Auricular Acupuncture (Experimental): Received true group auricular acupuncture twice weekly for a period of two months.
  Interventions: Other: True group auricular acupuncture
- Sham Group Auricular Acupuncture (Sham Comparator): Received sham group auricular acupuncture twice weekly for a period of two months.
  Interventions: Other: Sham group auricular acupuncture
- Wait-List Control Group (Other): Served as wait list control. Did not receive any acupuncture during the study period.
  Interventions: Other: Wait-List Control Group

INTERVENTIONS:
Other: True group auricular acupuncture — Received true group auricular acupuncture
  Arms: True Group Auricular Acupuncture
Other: Sham group auricular acupuncture — Received sham auricular acupuncture.
  Arms: Sham Group Auricular Acupuncture
Other: Wait-List Control Group — Received conventional care only. Eligible to receive true group auricular acupuncture once study period completed.
  Arms: Wait-List Control Group

SUMMARY:
The purpose of this study was to examine if group ear acupuncture improves Post-Traumatic Stress Disorder sleep difficulties among veterans who participated in Operations Enduring Freedom and Iraqi Freedom. This study also examined the degree of veteran acceptance for a group ear acupuncture procedure.

DETAILED DESCRIPTION:
Background: Approximately 70-91% of veterans with Post-Traumatic Stress Disorder (PTSD) report insomnia. Presently, conventional treatments for PTSD-related insomnia include medications, psychotherapy, and cognitive behavioral therapy. While some of these conventional treatments do improve PTSD-related insomnia, many of these treatments have limitations (e.g., medication effects, lengthy time commitments, psycho-social stigma). Because of these limitations, many veterans are increasingly turning to complementary and alternative therapies to relieve their symptoms. There is a growing body of research that shows that acupuncture may improve many health symptoms including depression, PTSD, addiction, headaches, musculoskeletal pain, and insomnia. However, to date, no study has specifically explored how acupuncture may affect PTSD-related insomnia. Because so many veterans with PTSD experience PTSD-related insomnia, and because the current conflicts in Southwest Asia are producing a new generation of combat veterans, it is critical that the VA explore innovative treatments for PTSD-related health concerns.

ELIGIBILITY:
Inclusion Criteria:

1. Combat veteran of Operation Iraqi Freedom or Operation Enduring Freedom conflicts;
2. Diagnosed with Post Traumatic Stress Disorder (PTSD) per Diagnostic Statistical Manual (DSM) IV criteria;
3. Have insomnia as indicated by a score equal to or greater than 8 on the Insomnia Severity Index (ISI);
4. Diagnosis of insomnia made after PTSD diagnosis; and
5. If on psychotropic medications, must be on stable psychotropic medication regimen for one month prior to enrollment in study.

Exclusion Criteria:

1. Does not speak English;
2. Not competent to sign informed consent;
3. History of moderate or severe traumatic brain injury
4. Start use of Continuous Positive Airway Pressure (CPAP) or Bilevel Positive Airway Pressure (BiPAP) during the study.
5. Experiencing severe psychiatric illness defined as suicidal ideation, homicidal ideation, or psychosis;
6. History of substance abuse Dependence (as defined per DSM IV criteria) during the one year preceding enrollment in the study OR history of illicit substance use for 3 months prior to study enrollment OR positive Audit C score at study enrollment (defined as score of 5 and above).
7. Received acupuncture during past 3 months.
8. On Coumadin, Heparin, or Lovenox
9. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-10; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Kennedy Prisco, MSN BC-ANP, Principal Investigator — Washington DC VA Medical Center, Washington, DC
Locations (1):
- Washington DC VA Medical Center, Washington, DC, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Letter, study flyers, and web sites were used to recruit Veterans to participate in this study at the Washington DC VA Medical Center. Veterans were recruited from November 2009 through June 2011.
Pre-assignment Details: Veterans who met initial telephone screening requirements were asked to participate in the full screening process. Of the 70 Veterans who provided informed consent, 35 Veterans were not randomized to study group because 1) did not meet full screening eligibility criteria; 2) did not complete baseline questionnaires; or 3) no longer eligible.
Groups:
- Sham Group Auricular Acupuncture: Received sham group auricular acupuncture.
- Wait-List Control Group: Served as wait-list control group. Did not receive any type of group ear acupuncture intervention--served as strict control and received conventional care only. Eligible to receive true group auricular acupuncture once study period was completed.
Period: Overall Study
Arm/Group | True Group Auricular Acupuncture | Sham Group Auricular Acupuncture | Wait-List Control Group
Started | 12 | 12 | 11
Completed | 8 | 8 | 9
Not Completed | 4 | 4 | 2
Not completed — Withdrawal by Subject | 3 | 3 | 2
Not completed — Protocol Violation | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: OEF/OIF Veterans with PTSD-related insomnia.
Groups:
- Wait List Control Group: Served as wait list control. Did not receive any acupuncture during the study period.
  Wait-List Control Group: Received conventional care only. Eligible to receive true group auricular acupuncture once study period completed.
- Total: Total of all reporting groups
Arm/Group | True Group Auricular Acupuncture | Sham Group Auricular Acupuncture | Wait List Control Group | Total
Number analyzed (Participants) | 12 | 12 | 11 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (11.4) | 37.9 (10.3) | 37.6 (8.0) | 37.8 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 4 | 10
  Male | 10 | 8 | 7 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 4 | 3 | 12
  White | 4 | 3 | 4 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 5 | 4 | 12
Post-Traumatic Stress Disorder Checklist-military version (PCL-M) [Mean (Standard Deviation); unit: units on a scale] — The Post-Traumatic Stress Disorder Checklist-military version (PCL-M) is a widely used, 17-item self-report measure of the 17 DSM-IV symptoms of PTSD. Items are rated on a 5-point Likert scale, and the total score (range 17-85) is obtained by summing the scores from each of the 17 items. Total scores of the PCL-M were reported, and higher scores indicate higher degrees of PTSD symptoms.
  units on a scale | 55.1 (11.4) | 57.8 (10.3) | 60.5 (14.4) | 57.9 (12.0)
PTSD symptom duration [Mean (Standard Deviation); unit: years] | 5.2 (3) | 6.3 (5.4) | 6.2 (3.2) | 5.9 (3.9)
PTSD-related insomnia duration [Mean (Standard Deviation); unit: years] | 4.9 (3) | 6.2 (5.6) | 5.7 (3.4) | 5.6 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: Perceived Sleep Quality
Description: Perceived sleep quality: subjective assessment of how restorative and undisturbed sleep has been. Measured by Insomnia Severity Index (ISI) and Morin sleep diary refreshness and soundness ratings.
  ISI: 7-item, self-report questionnaire based on DSM-IV criteria for insomnia. ISI scores range from 0 to 28 with higher scores reflecting greater insomnia. Total scores were reported, and an ISI cutoff total score of > 8 is indicative of probable insomnia.
  The Morin Sleep Diary refreshness and soundness ratings are based on a 5-point Likert scale with scores ranging from 1 to 5. Scores for these two questions were reported and higher scores indicate higher perceived sleep quality.
Time Frame: t=2 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | True Group Auricular Acupuncture | Sham Group Auricular Acupuncture | Wait List Control Group
Number analyzed (Participants) | 8 | 8 | 9
units on a scale
  Morin Sleep Diary Refreshness rating | 2.8 [2.1 to 3.4] | 2.6 [2.0 to 3.2] | 2.3 [1.8 to 2.9]
  Morin Sleep Diary Soundness Rating | 2.8 [2.1 to 3.4] | 2.8 [2.1 to 3.4] | 2.4 [1.8 to 3.1]
  Insomnia Severity Index total score | 16.3 [12.1 to 20.4] | 17.6 [13.5 to 21.7] | 20.1 [16.2 to 24]

2. Secondary Outcome: Fragmented Sleep Patterns-Total Sleep Time, Sleep Latency, and Naps
Description: Disruptive sleep patterns were analyzed by looking at Total Sleep Time (TST), Sleep Latency (SL), and Naps (short episodes of sleep at times other than bedtime). Morin sleep diaries (MSD) and wrist actigraphs (WA) were the study instruments used to collect this data.
Time Frame: t=2 months
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | True Group Auricular Acupuncture | Sham Group Auricular Acupuncture | Wait List Control Group
Number analyzed (Participants) | 8 | 8 | 9
minutes
  Total Sleep Time (TST)-MSD | 303.8 [242.8 to 364.7] | 397.3 [336.3 to 458.2] | 378.8 [321.3 to 436.2]
  Sleep Latency (SL)-MSD | 26.6 [6.4 to 46.9] | 31 [10.8 to 51.2] | 34.4 [15.4 to 53.5]
  Naps-MSD | 66.4 [31.9 to 100.9] | 16.9 [-17.6 to 51.4] | 15.9 [-16.7 to 48.4]
  Total Sleep Time (TST)-WA | 344.3 [288.3 to 400.2] | 407.6 [355.3 to 460.0] | 369.0 [316.7 to 421.3]
  Sleep Latency (SL)-WA | 22.6 [-2.5 to 47.6] | 34.1 [10.7 to 57.6] | 37 [13.6 to 60.4]
  Naps-WA | 33.9 [13.7 to 54] | 16.6 [-3.5 to 36.8] | 33.9 [13.7 to 54.0]

3. Secondary Outcome: Hypnotic Medication Use
Description: Amount of sleep medication taken by study participants. Measured by looking at demographic questionnaire results, chart reviews and Morin sleep diary (MSD).
Time Frame: t=2 months
Measure: Number; unit: participants
Arm/Group | True Group Auricular Acupuncture | Sham Group Auricular Acupuncture | Wait List Control Group
Number analyzed (Participants) | 8 | 8 | 9
participants
  Increased Hypnotic Medication Use | 0 | 1 | 0
  Decreased Hypnotic Medication Use | 1 | 0 | 0
  No Change | 2 | 3 | 3
  Not Applicable | 5 | 4 | 6

4. Secondary Outcome: Attrition Rates
Description: Examined attendance rates in attending group sessions to examine attrition rates.
Time Frame: t=2 months
Population: For this measure, participants in wait list control group not analyzed as did not participate in group sessions.
Measure: Mean (Standard Deviation); unit: % of sessions attended
Arm/Group | True Group Auricular Acupuncture | Sham Group Auricular Acupuncture | Wait List Control Group
Number analyzed (Participants) | 8 | 8 | 0
% of sessions attended | 68.0 (17.5) | 60.2 (21.2) |

5. Secondary Outcome: Number of Participants That Were Satisfied Based on Veteran Satisfaction Scores for True Group Acupuncture vs. Sham Group Acupuncture
Time Frame: t= 2 months
Population: For this measure, participants in wait list control group not analyzed as did not participate in group sessions.
Measure: Number; unit: participants
Arm/Group | True Group Auricular Acupuncture | Sham Group Auricular Acupuncture | Wait List Control Group
Number analyzed (Participants) | 8 | 8 | 0
participants
  Quality of Acupuncture (Very Good or Excellent) | 8 | 7 |
  Acupuncture addressed main health concern | 8 | 8 |

6. Secondary Outcome: Fragmented Sleep Patterns-Sleep Efficiency
Description: Disruptive sleep patterns that were analyzed by looking at Sleep Efficiency(SE). Morin sleep diaries (MSD) and wrist actigraphs (WA) were the study instruments used to collect this data.
Time Frame: t=2 months
Measure: Mean (95% Confidence Interval); unit: percentage of TST to time in bed
Arm/Group | True Group Auricular Acupuncture | Sham Group Auricular Acupuncture | Wait List Control Group
Number analyzed (Participants) | 8 | 8 | 9
percentage of TST to time in bed
  Sleep Efficiency (SE)-MSD | 77.3 [69.2 to 85.4] | 81 [72.9 to 89.1] | 80.8 [73.2 to 88.4]
  Sleep Efficiency (SE)-WA | 77.9 [70.4 to 85.3] | 83.1 [76.1 to 90] | 79.7 [72.7 to 86.7]

ADVERSE EVENTS:
Arm/Group | True Group Auricular Acupuncture | Sham Group Auricular Acupuncture | Wait List Control Group
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 0/12 | 1/12 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | True Group Auricular Acupuncture (N=12) | Sham Group Auricular Acupuncture (N=12) | Wait List Control Group (N=11)
Did not like acupuncture needles (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) — One participant in the sham auricular acupuncture group felt that the acupuncture needling was uncomfortable and as a result, did not wish to participate in study. The acupuncture needles were removed and no residual health effects were reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No